CLINICAL TRIAL: NCT00000810
Title: Randomized, Phase I/II, Dose-Ranging, Open-Label Trial of the Anti-HIV Activity of Delavirdine Mesylate (DLV; U-90,152S)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 260; 11237 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Delavirdine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Delavirdine mesylate
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
PRIMARY: To study the safety and tolerance of delavirdine mesylate ( U-90152 ) monotherapy. To compare the anti-HIV activity of three blood concentration levels of this agent with nucleoside analog monotherapy, either zidovudine ( AZT ) or didanosine ( ddI ), based on the reduction of HIV viral burden.

SECONDARY: To use pharmacokinetic parameters to assess the relationship between daily drug exposure and antiviral activity and toxicity of the U-90152, AZT, and ddI monotherapy. To assess anti-HIV activity using other disease markers.

Data suggest that bisheteroarylpiperazines (BHAPs) such as delavirdine mesylate are potent and safe anti-HIV agents and may have different biological behavior than other currently available non-nucleoside RT inhibitors.

DETAILED DESCRIPTION:
Data suggest that bisheteroarylpiperazines (BHAPs) such as delavirdine mesylate are potent and safe anti-HIV agents and may have different biological behavior than other currently available non-nucleoside RT inhibitors.

Patients are randomized to receive U-90152 at one of three doses (treatment arms I through III) or either AZT or ddI (treatment arm IV). Patients on arm IV who are AZT-naive receive AZT; those who are AZT-experienced receive ddI. Treatment continues for 24 weeks.

PER 12/22/94 AMENDMENT: All patients receiving U-90152 have the same starting dose, to attain one of three target trough levels.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* PCP prophylaxis.
* Topical antifungal agents, clotrimazole troches, nystatin oral suspension, topical ketoconazole, and oral fluconazole.
* Acyclovir (<= 1000 mg/day) as maintenance therapy for herpes simplex virus.
* Recombinant erythropoietin and G-CSF.
* Antibiotics for bacterial infections, unless specifically excluded.
* Symptomatic treatment such as antipyretics, analgesics, nonsteroidal anti-inflammatory agents, and antiemetics.
* Antacids.

Patients must have:

* HIV-1 infection.
* CD4 count 200 - 500 cells/mm3.
* Either no prior antiretroviral therapy or discontinued AZT monotherapy 3 or more weeks prior to study entry.

NOTE:

* Half of patients should be antiretroviral naive.

Prior Medication:

Allowed:

* Prior AZT.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancy other than minimal Kaposi's sarcoma.

Concurrent Medication:

Excluded:

* Rifabutin.
* Rifampin.
* Terfenadine.
* Astemizole.
* Loratadine.
* Trifluoperazine.
* Piperazine citrate.
* Any acute or chronic therapy for CMV, MAC, toxoplasmosis, or disseminated fungal infection.
* Non-study antiretroviral therapies, interferons, biologic response modifiers, and HIV vaccines.
* Systemic corticosteroids for more than 21 consecutive days.
* Foscarnet.
* Systemic cytotoxic chemotherapy for a malignancy.

Patients with the following prior conditions are excluded:

* History of pancreatitis (in patients who received prior AZT).
* History of grade 2 or worse peripheral neuropathy (in patients who received prior AZT).
* History of hypersensitivity to BHAP compounds (e.g., trifluoperazine - Stelazine, piperazine citrate - Antepar).

Prior Medication:

Excluded within 30 days prior to study entry:

* Any investigational medication.
* Interferon.
* Interleukin.
* Rifabutin.
* Rifampin.
* Terfenadine.
* Astemizole.
* Loratadine.
* Trifluoperazine.
* Piperazine citrate.

Excluded at any time:

* Prior ddI, ddC, d4T, or 3TC.
* Prior foscarnet.
* Prior BHAP compound or other non-nucleoside RT inhibitor.

Active substance abuse interfering with compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Study Completion 1996-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Para M, Study Chair; Fischl M, Study Chair
Locations (10):
- United States (10):
  - Stanford CRS, Stanford, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Howard University Hosp., Div. of Infectious Diseases, ACTU, Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Northwestern University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio

REFERENCES:
- [Background] Dereuddre-Bosquet N, Clayette P, Martin M, Fretier P, Jaccard P, Benveniste O, Lebeaut A, Dormont D. IL-10 and HIV-1 infection of human primary monocyte/macrophages. Int Conf AIDS. 1996 Jul 7-12;11(2):75 (abstract no WeA3107)
- [Background] Para M, Weinstock M. Retrospective analysis of protease inhibitor efficacy among patients failing a delavirdine regimen. Int Conf AIDS. 1998;12:59 (abstract no 12236)
- [Background] Morse G, Para M, Fischl M, Freimuth W. Concentration-targeted (CT) Delavirdine therapy in 82 patients in ACTG 260. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:118
- [Background] Para M, Morse G, Fischl M. Plasma protein binding of delavirdine in HIV-infected patients in ACTG 260. Int Conf AIDS. 1996 Jul 7-12;11(2):78 (abstract no WeB3131)
- [Background] Demeter L, Shafer R, Para M, Morse G, Freimuth W, Merigan T, Reichman R. Delavirdine (DLV) susceptibility of HIV-1 isolates obtained from patients (pts) receiving DLV monotherapy (ACTG 260). Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:113
- [Background] Para MF, Fischl M, Meehan P, Morse G, Wood K, Shafer R, Freimuth W, Demeter L, Holden-Wiltse J, Nevin T. ACTG 260: Randomized phase I/II concentration-controlled trial of the anti-HIV activity of delavirdine. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:163
- [Background] Demeter LM, Shafer RW, Meehan PM, Holden-Wiltse J, Fischl MA, Freimuth WW, Para MF, Reichman RC. Delavirdine susceptibilities and associated reverse transcriptase mutations in human immunodeficiency virus type 1 isolates from patients in a phase I/II trial of delavirdine monotherapy (ACTG 260). Antimicrob Agents Chemother. 2000 Mar;44(3):794-7. doi: 10.1128/AAC.44.3.794-797.2000. PMID 10681363
- [Background] Para MF, Meehan P, Holden-Wiltse J, Fischl M, Morse G, Shafer R, Demeter LM, Wood K, Nevin T, Virani-Ketter N, Freimuth WW. ACTG 260: a randomized, phase I-II, dose-ranging trial of the anti-human immunodeficiency virus activity of delavirdine monotherapy. The AIDS Clinical Trials Group Protocol 260 Team. Antimicrob Agents Chemother. 1999 Jun;43(6):1373-8. doi: 10.1128/AAC.43.6.1373. PMID 10348755